CLINICAL TRIAL: NCT00235859
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase III Study of the Human Anti-TNF Antibody Adalimumab Administered as Subcutaneous Injections in Korean Rheumatoid Arthritis Subjects Treated With Methotrexate
Brief Title: Adalimumab Administered in Korean Rheumatoid Arthritis Subjects Treated With Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Eisai Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M02-556
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; adalimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: adalimumab
Drug: methotrexate

SUMMARY:
The purpose of the study is to assess the safety and efficacy of adalimumab compared to placebo in subjects with rheumatoid arthritis on methotrexate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Meet ACR criteria for diagnosis of active RA and have at >6 swollen joints and >9 tender joints
* Subjects must have received at least one prior DMARD besides MTX, but may have had efficacy failures on no more than four standard DMARDs other than MTX
* Therapy with MTX for at least 6 months prior to screening and on a stable dose of MTX for at least 4 weeks prior to screening visit
* Age 18 years and older

Exclusion Criteria:

* Prior treatment with any TNF antagonist, including adalimumab
* History of clinically significant drug or alcohol abuse in the previous year, iv drug abuse, active infection with listeria or tuberculosis (TB), lymphoma or leukemia,and any malignancy with the exception of successfully treated non-metastatic basal-cell carcinoma of the skin.
* Subjects may not have been administered a live vaccine within three months prior to study drug administration or during the study, treatment with any other investigational agent within 30 days or 5 half-lives of the agent, whichever is longer, prior to the screening evaluation, treatment with any investigational biologic agent, including anti-CD4 antibody, within 6 months prior to the screening evaluation, prior treatment with any TNF antagonist, including Adalimumab, prior exposure to alkylating agents such as chlorambucil or cyclophosphamide.
* Chest X-ray with calcified granuloma and/or pleural scarring
* Positive TB skin test, RT23 dose skin test, >5 mm at 48 to 72 hours
* Unstable ischemic heart disease, active inflammatory bowel disease, active peptic ulcer disease, recent stroke (within 3 months of the screening evaluation) or any poorly controlled medical condition
* Intra-articular, intramuscular or iv administration of corticosteroids within 4 weeks prior to screening evaluation
* Female who is pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2003-07

PRIMARY OUTCOMES:
ACR20

SECONDARY OUTCOMES:
Safety parameters

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Paperiello, Study Director — Abbott

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778